CLINICAL TRIAL: NCT00286390
Title: Outcomes and Cost Assessment of Acupuncture in the Treatment (OCAT) of Pain Patients at Malcolm Grow USAF Medical Center
Brief Title: Acupuncture for Acute and Chronic Pain in Air Force Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: CRO-04-01; FMG2005-0002H
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this project is to conduct a scientifically rigorous investigation of the clinical outcomes, quality of life, and cost associated with the delivery of acupuncture in the treatment of acute and chronic pain in patients at Malcolm Grow Medical Center, Andrews Air Force Base.

The specific aims of this study are to:

1. Gather outcomes and patient satisfaction data on patients receiving acupuncture treatment for acute and chronic pain.
2. Perform an analysis of costs, including any system cost savings, associated with providing acupuncture services to pain patients.
3. Serve as a model to expand the project to Scott AFB and Travis AFB as per the request of the Air Mobility Command Surgeon General. (AMC/SG).

DETAILED DESCRIPTION:
Adult patients referred to the MGMC Acupuncture Clinic for this study must have an established Western medical diagnosis, have exhausted all standards of care for the reduction and/or resolution of pain, meet the inclusion and exclusion criteria and be clinically evaluated prior to entry in the study. 1000 patients will be entered into the study; no male and female patient ratios will be required. Patients under 18 years of age will be excluded. There are no upper age limits.

Acupuncture point(s) selection and acupuncture techniques will be individualized for each patient. All treatments will be approved by the physician principal investigator. Treatment will generally be administered with the patient either prone, supine, or seated position. Standards of reporting interventions in controlled trials of acupuncture, based on STRICTA requirements, will be followed. The following acupuncture data will be collected:

* Acupuncture point locations (palpation or electronic detection)
* Techniques employed: (e.g. dry needling, acupuncture, electro-acupuncture , auriculotherapy, electro-auriculotherapy, laser, piezo-electrical stimulation micro-current techniques, E-field)
* Types of needles employed (e.g. ASP gold/stainless steel, needle tacks, Seirin needles, etc.)

Baseline demographic data and information on pain levels (using the Numerical Rating Scale), patient satisfaction (using the Patient Satisfaction Questionnaire), functional health status (using the SF-8), and concomitant medical care (including medication use) will be collected prior to treatment. Follow-up data on pain levels and concomitant medical care will be collected via telephone 24 hours, 1 week, 2 weeks, and 4 weeks post-therapy. Patient satisfaction and functional health status data will be collecetd again at 4 weeks post-treatment. Relapses of pain will be noted and appropriately evaluated. In addition, the following clinical data will be collected:

* Subjective, Objective, Assessment, and Treatment(SOAP) parameters
* Medication use
* Range of motion

A cost analysis will be performed by comparing patients who seek acupuncture treatment to those who receive only conventional medical care during the same time period, by matching cohorts based on ICD-9 diagnostic codes and basic demographic information.

A series of appropriate parametric and nonparametric tests will be performed to look for pre-post differences in patient outcomes on a number of relevant baseline variables; including demographic information, intensity and duration of pain, SF-8 scores, patient satisfaction, and utilization of concomitant medical services.

An ancillary study will be conducted to investigate personality factors and pretreatment expectations as predictors of treatment outcome of medical acupuncture. Specific Aims of this ancillary study include:

1. To assess perceived health outcomes after acupuncture treatment by military medical acupuncturists.
2. To identify psychosocial and demographic predictors of perceived health outcomes from acupuncture treatment by military medical acupuncturists.
3. To help clarify which patients are more likely to respond to acupuncture and hence more likely to benefit from a referral to a trained medical acupuncturist.

ELIGIBILITY:
Inclusion Criteria:

* Western diagnosis of acute or chronic pain syndromes
* Previously treated western standard of care
* Written Informed Consent
* Over the age of 18

Exclusion Criteria:

* Unwilling or unable to participate in study treatment and follow-up
* Unable to give informed consent for any reason
* Allergic reaction to adhesive tape, gold or other components of the acupuncture needles
* Pregnancy
* Pacemaker
* Electronic stimulator of any sort
* Herbal preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-03; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Level of Pain at Conclusion of Study, as measured by using a 0-10 Numerical Rating Scale (NRS) | Baseline; Final assessment

SECONDARY OUTCOMES:
Pain Level, as measured by using a 0-10 Numerical Rating Scale (NRS) and Medication Use | Baseline; Immediately after tx; 24 hours after tx

CONTACTS AND LOCATIONS:
Overall Officials: COL Richard C Niemtzow, MD, PhD, MPH, Principal Investigator — United States Air Force
Locations (1):
- Malcolm Grow Medical Center (MGMC), Andrews Air Force Base, Andrews Air Force Base Census Designated Place, Maryland, United States